CLINICAL TRIAL: NCT02838966
Title: Preoperative Nutritional Supplementation With Immunomodulators for Patients With Resectable Pancreatic Adenocarcinoma: Efficacy and Optimal Dose
Brief Title: Preoperative Nutrition With Immune Enhancing Nutritional Supplement (Immunomodulation)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor did not want to supply further product
Sponsor: University of Louisville (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Prejesh Philips, Assistant Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Immunonutrition PDAC #14-0779
Record Dates: First submitted 2015-11-18; First posted 2016-07-20 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: immunomodulation; immunonutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nestle IMPACT Advanced Recovery 1 (Active Comparator): 1 can per day for 5 days prior to surgery
  Interventions: Dietary Supplement: Nestle IMPACT Advanced Recovery
- Nestle IMPACT Advanced Recovery 2 (Active Comparator): 2 cans per day for 5 days prior to surgery
  Interventions: Dietary Supplement: Nestle IMPACT Advanced Recovery
- Nestle IMPACT Advanced Recovery 3 (Active Comparator): 3 cans per day for 5 days prior to surgery
  Interventions: Dietary Supplement: Nestle IMPACT Advanced Recovery
- Nestle Boost High Protein Drink - Control Arm (Active Comparator): 4 cans per day for 5 days prior to surgery
  Interventions: Dietary Supplement: Nestle Boost High Protein Drink

INTERVENTIONS:
Dietary Supplement: Nestle IMPACT Advanced Recovery
  Arms: Nestle IMPACT Advanced Recovery 1; Nestle IMPACT Advanced Recovery 2; Nestle IMPACT Advanced Recovery 3
Dietary Supplement: Nestle Boost High Protein Drink
  Arms: Nestle Boost High Protein Drink - Control Arm

SUMMARY:
The purpose of this study is to determine the optimal effective dose for preoperative nutritional supplementation with immunomodulators on immune function and perioperative outcomes following pancreaticoduodenectomy for pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Study Objectives: The primary objective of this study is to determine the optimal effective dose for preoperative nutritional supplementation with immunomodulators on immune function and perioperative outcomes following pancreaticoduodenectomy for pancreatic adenocarcinoma.

Primary Endpoints:

The primary endpoints will be effect on immunological profile (circulating Myeloid derived suppressor cells, circulating B cells, NK cells, CD4 and CD8 cells), serum arginine levels, immunological milieu of the tumor (tumor infiltrating lymphocytes), overall morbidity rate and infectious complication rates.

Secondary Endpoints:

* Monitor Safety and Tolerability
* Hospital Length of Stay
* Readmission rate
* One-year event free survival
* Effect on nutritional parameters (serum total protein, prealbumin, albumin and transferrin)
* Effect on acute phase reactants (CRP, IL6, TNF alpha)

Study Design: This is a 1:1:1:1 four-arm single center prospective randomized feasibility study to compare preoperative nutritional supplementation with an enhanced formula containing immune-modulating agents (IMPACT AR) for 5 days with 1,2 or 3 cans versus 5 days of 3 cans of comparable iso-caloric iso-nitrogenous supplementation (Boost) for patients with resectable pancreatic adenocarcinoma.

Number of Patients 20 (5 in each arm) Eligibility Criteria: Patients over 18 years of age, who have histologic and/or radiologic evidence of pancreatic adenocarcinoma in the head of the pancreas, who have been deemed resectable, and who are able to give informed consent, will be eligible Exclusion criteria would include Active uncontrolled bacterial, viral or fungal infection within 21 days of study entry OR Inability to take oral, nasojejunal or jejunostomy tube nutritional supplements OR patients on chronic steroid therapy (i.e. greater than 3 months)

Nutritional Supplement interventions:

Patients randomized to the TEST intervention will receive Impact Advanced Recovery™ formula, which is a commercially available oral nutrition supplement drink that is supplied in 237mL containers. Each serving provides 1.4 kcal/mL (340 kcal/serving) of which 22% of the kcal are derived from protein (18.1 gm protein/serving), in addition to their regular diet. Patients randomized to CONTROL Boost® High Protein Drink will consume their regular diet and 4 cans of Boost per day for 5 days preoperatively (to maintain equivalent supplementation in terms of calories and protein with the group receiving the highest dose of Impact AR).

Study procedure:

Screening/baseline assessments will performed prior to the first treatment within approximately four weeks of the treatment and will include a detailed medical history and physical examination,standard of Care Laboratory tests (CBC, CMP), tumor markers: as indicated: CEA and CA19-9; and coagulation (baseline and as clinically indicated): INR, PTT, PT. Imaging to confirm respectability would include a high quality tri-phasic CT scan with 0.7mm cuts or Dynamic MRI with contrast to confirm the absence of metastatic disease Study specific tests include pre-treatment and post treatment (Office visit/ pre-anesthesia visit, Morning of surgery, postop day 5)

* Nutritional parameters and acute phase reactants: serum prealbumin, albumin, transferrin, CRP, IL6, TNF alpha
* Serum arginine,
* MSDC (myeloid derived suppressor cell) assay of fresh blood and Arginase I expression Study procedure at the time of surgery: Semi-quantitative assay of Tumor infiltrating lymphocytes from tissue block of tumor obtained at time of surgery. Tumor tissue will also be banked for post hoc tests if needed.

During follow up visits history and physical examination, performance Status evaluation and Standard of care Laboratory Tests (CBC, CMP, and Tumor Marker Assessment as clinically indicated per the discretion of the investigator would be done approximately every three months). Imaging during follow up include a CT/MRI for disease status (approximately every three months during follow-up) Adverse Event Monitoring and Concomitant Medication monitoring will be done out to 90 days

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, of any race or sex, with histologic and/or radiologic proof of pancreatic adenocarcinoma (PDAC)
* PDAC that is deemed resectable by the operating surgeon
* Non-pregnant with an acceptable contraception method in premenopausal women
* Signed, written informed consent

Exclusion Criteria:

* Active bacterial, viral or fungal infection within 21 days of study entry
* Women who are pregnant or breast feeding
* Evidence of metastatic disease
* Presence of another malignancy with the exception of cervical carcinoma in situ and stage I basal or squamous cell carcinoma of the skin
* Inability to take oral or nasojejunal nutritional supplements
* Patients with immunodeficiency conditions
* Patients on chronic steroid therapy
* Patients with know sensitivity to arginine, omega-3 fatty acids or glutamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Change in levels of circulating Myeloid derived suppressor cells | Within 2 weeks of study intervention (at pre-anesthesia visit) to surgery. Study intervention to start 5 days before surgery
  The variable that will be compared in this analysis will be
  • Change in circulating Myeloid derived suppressor cells before and after intervention (before intervention: within 2 weeks before surgery; after intervention: day of surgery)
Overall morbidity rate. | 30 day morbidity from surgery
  The variables that will be compared in this analysis will be
  • overall morbidity rate (adverse effects): number of patients with adverse effects and total number of adverse effects as assessed by CTCAE v4.0 (which includes number of patients with serious adverse effects: Grade 3 or higher, CTCAE v4.0 and number of patients with infectious complication rates)

SECONDARY OUTCOMES:
Tolerability of Supplement | 90 days from surgery
  Tolerability of supplement: as defined as ability to complete the nutritional intervention using a patient log.
Hospital length of stay | 90 days from surgery
  Length of hospital stay (in days)
Change in serum arginine levels | Within 2 weeks of study intervention (at pre-anesthesia visit) to surgery. Study intervention to start 5 days before surgery
  Arginine level assay

CONTACTS AND LOCATIONS:
Overall Officials: Prejesh Philips, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States